CLINICAL TRIAL: NCT01843049
Title: Dose Escalation Using a Simultaneous Integrated Boost Technique Based on 18FDG-PET/CT for Unresectable Thoracic Esophageal Cancer: a Phase I/II Trial
Brief Title: Dose Escalation by Boosting Radiation Dose Within the Primary Tumor Using 18FDG-PET/CT for Unresectable Thoracic Esophageal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaolong Fu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013ESO_FU_01
Record Dates: First submitted 2013-04-24; First posted 2013-04-30 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiotherapy+chemotherapy (Experimental): Radiotherapy:
  LEVEL 1: dose given at PTV-G and PTV-C will be 64Gy/32 fractions and 50Gy/25 fractions.
  LEVEL 2: dose given at PTV-G and PTV-C will be 63Gy/28 fractions and 50.4Gy/28 fractions.
  LEVEL 3: dose given at PTV-GR (with an integrated boost to the 50% SUVmax area of the primary tumor of the pre-treatment 18FDG-PET/CT scan), PTV-G and PTV-C will be 70Gy/28 fractions, 63Gy/28 fractions and 50.4Gy/28 fractions.
  LEVEL 4: dose given at PTV-GR (with an integrated boost to the 50% SUVmax area of the primary tumor of the pre-treatment 18FDG-PET/CT scan), PTV-G and PTV-C will be 70Gy/25 fractions, 62.5Gy/25 fractions and 50Gy/25 fractions.
  Chemotherapy:
  Concurrent chemotherapy: Cisplatin 25mg/m2 IV daily on Days 1-3 and 29-31 plus 5-FU 500mg/m2 IV continuous infusion over 24 hours daily on Days 1-4 and 29-32.
  Consolidation chemotherapy: Cisplatin 25mg/m2 IV daily on Days 1-3 plus 5-FU 600mg/m2 IV daily on Days 1-5, cycled every 4 weeks for 2 cycles.
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapy (5-FU+DDP)

INTERVENTIONS:
Radiation: Radiotherapy — Patients will receive from 5 to 6 weeks 5 days a week radiations. The dose of radiation will depend on the level they will be included.
Drug: Chemotherapy (5-FU+DDP) — Patients will receive 2 cycles of concurrent chemotherapy (cisplatin 25mg/m2 IV daily on Days 1-3 and 29-31 plus 5-FU 500mg/m2 IV continuous infusion over 24h daily on Days 1-4 and 29-32) during radiotherapy period. Consolidation chemotherapy (cisplatin 25mg/m2 IV daily on Days 1-3 plus 5-FU 600mg/m2 IV daily on Days 1-5, cycled every 4 weeks) will be given for 2 cycles one month after the end of radiochemotherapy.

SUMMARY:
Most local failures after definitive chemoradiation for unresectable esophageal cancer occur in the gross tumor volume (GTV). And the metabolic active areas post-treatment were located in the high FDG uptake areas prior to the radiotherapy. The hypothesis is that selective dose boost to the esophageal GTV could be safely delivered using a simultaneous integrated boost (SIB) technique, and that boosting the high 18F-deoxyglucose (FDG) uptake areas of the esophageal GTV defined prior to treatment may improve local tumor control.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven diagnosis of esophageal squamous cell carcinoma.
2. ECOG performance status 0-1.
3. Able to swallow semifluid diet.
4. Patients must not have received either radiotherapy or chemotherapy.
5. Technically unresectable, medically inoperable, or surgery declined by the patient.
6. SUVmax in the pre-treatment FDG-PET scan > 5 for the primary tumor and the length of the primary tumor ≤10cm.
7. Normal liver and renal function and adequate bone marrow reservation.
8. Meet the requirements of the dose limitation to the critical organ: V20≤25%，Dmean≤15Gy for lung; Dmax ≤45Gy for spinal cord，Dmean ≤20Gy for liver.
9. Written, signed informed consent.

Exclusion Criteria:

1. Other malignancy histology.
2. Any evidence of visceral metastases.
3. Prior radiotherapy to the thorax or systemic therapy for esophageal cancer.
4. Evidence of deep esophageal ulcer or esophageal perforation.
5. Weight loss ≥10% within half year or cachexia.
6. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ.
7. History of cardiac disease: congestive heart failure > NYHA class 2, active CAD, cardiac arrythmias requiring anti-arrhythmic therapy or uncontrolled hypertension within the last 12 months.
8. Concurrent uncontrolled medical conditions.
9. Pregnant or lactating women.
10. Drug addiction, alcoholism or AIDS.
11. Uncontrolled seizures or psychiatric, behavioural disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity(DLT) | 3 months after the finish of the radiotherapy

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
Progression-free survival (PFS) | 3 years
Failure patterns | 3 years
Late toxicity | 3 years
  Esophageal perforation, esophageal bleeding or late radiation-induced lung or heart injury of grade 3 or above(CTCAE3.0)

OTHER OUTCOMES:
Local recurrent rate within the >50% SUVmax region of the primary tumor | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Fu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Yu W, Cai XW, Liu Q, Zhu ZF, Feng W, Zhang Q, Zhang YJ, Yao ZF, Fu XL. Safety of dose escalation by simultaneous integrated boosting radiation dose within the primary tumor guided by (18)FDG-PET/CT for esophageal cancer. Radiother Oncol. 2015 Feb;114(2):195-200. doi: 10.1016/j.radonc.2014.12.007. Epub 2015 Jan 10. PMID 25586952